CLINICAL TRIAL: NCT06749353
Title: Distraction Manuever to Reduce Intraoperative Anxiety During Vasectomy Procedure Under Local Anesthesia
Brief Title: Virtual Reality to Reduce Intraoperative Anxiety in Vasectomies Under Local Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P/23-079/
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: anxiety; biomarkers; cortisol; vasectomy; virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: PRE POST INTERVENTION STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- USUAL (No Intervention): In the control group, we will perform the surgical procedure as usual, without any distraction maneuvers, under local anesthesia.
- VIRTUAL REALITY (Experimental): In the study group, we will perform the vasectomy under local anesthesia and provide patients with virtual reality glasses as a distraction technique, aiming to reduce intraoperative anxiety.
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — We will use a virtual reality glasses with the 'Lending Moments' program, where patients can experience a sunset on a paradise beach while listening to a soothing voice that guides them through the experience with relaxation and meditation techniques. During this time, we will proceed with the surgical intervention.
  Arms: VIRTUAL REALITY

SUMMARY:
Vasectomy is an elective and ambulatory surgery, typically performed under local anaesthesia. The most common problem that we have found among patients is the anxiety and the apprehension to face the procedure.

Virtual reality (VR), as a novel tool, is relatively underutilized in such medical context. It has been successfully employed across various medical domains, aiding in the training of surgeons, enhancing procedural planning, and offering psychological support to patients.

This project aims to assess the effectiveness of employing distraction maneuverers, using virtual reality glasses, during the intraoperative period on vasectomy surgery, to mitigate anxiety during the surgical process.

We want to develop a randomized clinical trial, single-centre study with a control group (conventional procedure) and an intervention group (Virtual reality Glasses). Anxiety was measured using cortisol level through a biomarker saliva test, involving pre and post-procedure samples for each patient. Additionally, we used the State-Trait Anxiety Inventory (STAI) pre and post procedure to evaluate the anxiety and the correlation with the cortisol levels, To evaluate the patient's satisfaction with the used of VR glasses a satisfaction survey was developed. The study protocol has received approval from the ethical committee of our institution.

The investigators expect to find statistically significant differences in salivary cortisol levels on postoperative samples to prove that VR helps to have a better experience and reduce the intraoperative anxiety.

DETAILED DESCRIPTION:
Upon arrival at the ambulatory surgery unit (ASU) for a vasectomy, the patient will be informed about the study. If they agree to participate, they will be given an informed consent form to read and sign.

At the ASU, the nurse will record the patient's age and provide the STAI Trait-State scale for completion before entering the operating room. A preoperative saliva sample will be collected to analyze cortisol levels. The patient will be entered into the database and randomized into either the control or intervention group.

Once in the operating room, the patient will be positioned, and a preoperative verification will be performed. The urologist will speak with the patient to provide information, explain the surgery, and confirm the procedure. Heart rate and blood pressure will be recorded. For patients in the intervention group, virtual reality glasses with the "Lending Moments" program will be applied. This program simulates a sunset on a paradisiacal beach while a calming voice guides the patient through relaxation and meditation techniques. The surgical procedure will be performed during this time. Heart rate and blood pressure will be recorded again during the procedure.

Upon completion of the surgery, the patient will be informed and the virtual reality glasses will be removed for patients in the intervention group. The patient will be accompanied to the waiting room, where a postoperative saliva sample will be collected. The patient will be given the STAI State scale and a questionnaire to assess their experience. Heart rate and blood pressure will be recorded postoperatively.

Samples will be sent to the laboratory for processing the same day. Descriptive statistics will be computed, including means (with standard deviations), frequencies, and proportions, according to the variable type at each phase. The Kolmogorov-Smirnov test will be used to assess the normality of quantitative variables. For variables that do not follow a normal distribution, medians (and the 25th and 75th percentiles) will be reported.

For bivariate analysis, Student's t-test or the Mann-Whitney U test will be used for quantitative variables, and the chi-squared test will be used for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 20 and 90 years old
* Intervention between 8 am to 12 am.
* Vasectomy under local anesthesia

Exclusion Criteria:

* Language barrier
* Oncological urological syurgery
* Surgery time superior to 30 minuts
* Intellectual disability
* STAI Trait > 70%
* Intervention after 12 am

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biomarker | 96 weeks
  Cortisol is a commun stress biomarker used in many studies.
Psicological Scale | 96 weeks
  We will mesure the intraoperative anxiety

SECONDARY OUTCOMES:
Patient experience | 96 weeks
  The patient will complete a questionnaire regardind the attention recieved and subjective anxiety percieved. It has 9 questions, where the patient could evaluate the experience lived during the surgery from 1, being a very bad experience, to 10 being better experience possible.
Blood preasure | 96 weeks
Heart rate | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olga Monistrol, RN, MsC, PhD, Principal Investigator
Locations (1):
- Hospital Univesitari Mútua de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (1) Mallari B, Spaeth EK, Goh HX, Slijepcevic N, Guo Y, Doherty CJ, Yeomans DC, Burns LC. Virtual Reality Distraction for Pain Control During Medical Procedures: A Systematic Review of Randomized Controlled Trials. Clin J Pain. 2019